CLINICAL TRIAL: NCT05066802
Title: A Phase 2 Trial of Neoadjuvant Modified FOLFIRINOX Chemotherapy for Resectable Pancreatic Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0485
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Resectable Pancreatic Adenocarcinoma
Keywords: resectable pancreatic cancer; Neoadjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- modified FOLFIRINOX (Experimental): oxaliplatin 85 mg/m2 D1 + leucovorin 400mg/m2 D1 + irinotecan 150 mg/m2 D1 + 5-FU 2,000 mg/m2 42~46h continuous infusion, every other week for 6 cycles (12 weeks).
  Interventions: Drug: neoadjuvant modified FOLFIRINOX

INTERVENTIONS:
Drug: neoadjuvant modified FOLFIRINOX — oxaliplatin 85 mg/m2 D1 + leucovorin 400mg/m2 D1 + irinotecan 150 mg/m2 D1 + 5-FU 2,000 mg/m2 42~46h continuous infusion, every other week for 6 cycles (12 weeks) before surgery.

SUMMARY:
Within the next decade, pancreatic ductal adenocarcinoma (PDAC) is expected to rise to the second leading cause of cancer-related mortality. To increase the survival, various peri-operative treatments have been tested, and adjuvant FOLFIRINOX or gemcitabine plus capecitabine is now standard of care after surgical resection for localized PDAC. Even with superior survival among various disease extent of PDAC, resectable PDAC still shows poor outcomes with surgery followed by adjuvant chemotherapy. This phase II study is investigating the role of modified-FOLFIRINOX as neoadjuvant treatment for resectable PDAC.

DETAILED DESCRIPTION:
This phase II study is designed to evaluate the efficacy and safety of modified FOLFIRINOX as neoadjuvant treatment for resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pancreatic ductal adenocarcinoma confirmed by histological or cytopathological examination
2. Pancreatic adenocarcinoma patients evaluated as resectable according to the following criteria in imaging tests including CT or MRI (NCCN guideline criteria, if all of the following criteria are satisfied) A. No tumor contact with the major arterial structures of the Celiac axis [CA], superior mesenteric artery [SMA], and common hepatic artery [CHA].

   B. When there is no contact between the tumor and the major vein of the superior mesenteric vein (SMV) or portal vein (PV), or within 180° even if there is contact, and there is no venous atypicality.
3. Patients who have not undergone surgical resection and systemic chemotherapy for pancreatic cancer.
4. Patients whose ECOG activity ability index is 0 to 1
5. Patients who are willing and able to provide written informed consent for this study.
6. Patients over the age of 19 at the time of signing the subject consent form.
7. Patients with evaluable lesions according to RECIST 1.1.
8. Patients with adequate organ function.

Exclusion Criteria:

1. Histologic diagnosis other than pancreatic ductal adenocarcinoma (eg, neuroendocrine tumor, etc.)
2. Patients with distant metastases including central nervous system (CNS) metastases or peritoneal metastases
3. Patients with moderate acute or chronic medical conditions or abnormal findings on examination, which are judged to affect the results of this study
4. Patients who have participated in a study in which investigational drugs are used and are currently receiving investigational drugs or used investigational drugs or medical devices within 4 weeks prior to the first administration of this investigational drug.
5. Those who received chemotherapy, targeted small molecule agents, or radiotherapy within 2 weeks prior to Day 1 of the study, or who have not yet recovered (Grade 1 or lower or baseline level) from adverse reactions due to previously administered drugs patient.
6. Patients with known aggravation within the past 3 years or other malignant tumors requiring active treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | Post surgery (within one week)
  R0 resection rate with pathology report after curative aim surgery.

SECONDARY OUTCOMES:
overall survival | up to 2 years
  overall survival is defined as time interval from cycle 1 day 1 to tumor death/last follow-up.
Progression Free Survival | up to 2 years
  Progression Free Survival is defined as time interval from cycle 1 day 1 to tumor progression/death/last follow-up
disease-free survival | up to 2 years
  disease-free survival is defined as time interval from operation day to tumor progression/death/last follow-up
Objective response rate | 3 months
  Objective response rate is defined as rate of patients with complete remission (CR) or partial remission (PR) based on RESIST1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Choong-kun Lee, Principal Investigator — Division of Medical Oncology, Yonsei Cancer Center, Yonsei Univ. College of Medicine, Korea
Locations (1):
- Division of Medical Oncology, Yonsei Cancer Center, Yonsei Univ. College of Medicine, Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No